CLINICAL TRIAL: NCT01012700
Title: A Randomized, Placebo-controlled, Phase I Study to Evaluate the Safety and Immunogenicity of Poly ICLC (Hiltonol) in Healthy Volunteers
Brief Title: Study to Evaluate the Safety and Immunogenicity of Poly ICLC (Hiltonol) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: MAC-0682
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — poly ICLC

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- intranasal or IV (No Intervention): Each study group consists of 12 volunteers randomized in a 2:1 ratio to receive poly ICLC or placebo: in group 1, 8 volunteers will be administered poly ICLC and 4 volunteers will be administered placebo, subcutaneously; and in group 2, 8 volunteers will be administered poly ICLC and 4 volunteers will be administered placebo, intranasally. A total of up to 24 volunteers will be enrolled in the study.
- Hiltonol (poly ICLC) (Active Comparator): Each study group consists of 12 volunteers randomized in a 2:1 ratio to receive poly ICLC or placebo: in group 1, 8 volunteers will be administered poly ICLC and 4 volunteers will be administered placebo, subcutaneously; and in group 2, 8 volunteers will be administered poly ICLC and 4 volunteers will be administered placebo, intranasally. A total of up to 24 volunteers will be enrolled in the study.
  Interventions: Drug: Hiltonol (poly ICLC)

INTERVENTIONS:
Drug: Hiltonol (poly ICLC) — 2 mg administered subcutaneously or intranasally to healthy volunteers
  Arms: Hiltonol (poly ICLC)

SUMMARY:
Vaccines induce protective immunity against numerous infectious diseases. However, current vaccines have limited efficacy against challenging infections like tuberculosis, malaria and HIV. Protein vaccines are safe but, typically, they induce weak T cell immunity when administered alone. Therefore, special attention is being given to adjuvants, which are enhancers of immunity, that mature antigen presenting immunostimulatory dendritic cells (DCs). Our goal is to study in humans the mechanism whereby synthetic adjuvants, acting on defined pattern recognition receptors (PRR), enhance T and B cell immunity. In preclinical studies, the investigators' laboratory has found in mice that poly IC and its analog poly ICLC are superior adjuvants for T cell mediated immunity relative to other agonists for PRR. In this study the investigators propose to study the safety and the innate immune responses to poly ICLC in multiple blood cell types, including three different subsets of DCs when administered subcutaneously or intranasally to healthy volunteers. Poly ICLC is a stabilized double stranded RNA which has been extensively studied in humans with a favorable safety profile.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males and females, as assessed by a medical history, physical exam, and laboratory tests
2. Age of at least 18 years on the day of screening and no greater than 60 years at time of drug/placebo administration
3. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study (screening plus 4 weeks)
4. In the opinion of the principal investigator or designee, has understood the information provided. Written informed consent needs to be given before any study-related procedures are performed
5. Willing to undergo HIV testing and counseling, and receive HIV test results
6. If a sexually active male, willing to use an effective method of contraception (condoms, anatomical sterility) throughout the study period and will be advised not to get his partner pregnant for 6 weeks after study drug administration
7. Females of child-bearing potential must agree to use one of the following methods of contraception for 2 weeks prior to date of screening evaluation through 6 weeks after study drug administration:

   * Be surgically sterile Be abstinent (or willing to be)
   * Use oral contraceptives, or other form of hormonal birth control including hormonal vaginal rings or transdermal patches
   * Use an intra-uterine device (IUD)
   * Use (by ensuring her male partner(s) uses) barrier contraception (condom) with spermicide
   * Any other equivalent (as judged by the investigative team) methods of contraception

Exclusion Criteria:

1. Any clinically significant abnormality on history or examination including history of immunodeficiency or autoimmune disease; use of systemic corticosteroids, immunosuppressive, anticancer, or other medications considered significant by the trial physician within the last 6 months
2. Confirmed HIV-1 or HIV-2 infection
3. A medical history that includes any chronic medical problem that requires daily topical nasal medications, prior nasal or sinus surgery (including trans-nasal approaches of other organs such as pituitary, allergic rhinitis, chronic sinusitis, or any other nasal inflammatory disease that requires daily intranasal or oral medication)
4. A medical history that includes any chronic pulmonary conditions including but not limited to asthma, chronic obstructive pulmonary disease and chronic bronchitis
5. Any clinically significant acute or chronic medical conditions requiring care of a physician (e.g., diabetes, coronary artery disease, rheumatologic illness, malignancy, substance abuse) that in the opinion of the investigator would preclude participation
6. Any laboratory value outside of reference range, with the exception of any non-clinically significant Grade 1 elevations of liver function tests (AST, ALT, direct/total bilirubin), CBC, as determined by the Principal Investigator or her designee
7. Confirmed diagnosis of hepatitis B (surface antigen, HbsAg); hepatitis C (HCV antibodies) or active syphilis
8. If female, pregnant, planning a pregnancy during the trial period or lactating
9. Receipt of a live attenuated vaccine within 30 days or other vaccine within 14 days of poly ICLC administration
10. Receipt of blood transfusion or blood products 6 months prior to drug administration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of a single dose of 2mg of poly ICLC (Hiltonol) administered to healthy volunteers. | 12 months

SECONDARY OUTCOMES:
To evaluate the innate immune responses to poly ICLC in multiple blood cell types in addition to whole PBMCs and three different subsets of dendritic cells after administration to healthy volunteers at different timepoints of administration. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marina Caskey, MD, Principal Investigator — Instructor in Clinical Investigation
Locations (1):
- The Rockefeller University, New York, New York, United States